CLINICAL TRIAL: NCT03191526
Title: A Phase 3 Multicenter, Randomized, Double-Blind and Placebo-Controlled Study, and Open Study of KW-0761 in Patients With HTLV-1 Associated Myelopathy (HAM)
Brief Title: A Study of KW-0761 in Subjects With HTLV-1 Associated Myelopathy (HAM)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to not achieving the primary outcome.
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0761HAM-001
Record Dates: First submitted 2017-06-13; First posted 2017-06-19 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: HTLV-1 Associated Myelopathy
MeSH Terms: conditions — Paraparesis, Tropical Spastic | interventions — mogamulizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KW-0761 0.3 mg/kg IV (Experimental): Intravenous injection every 12 weeks. Duration of double-blind treatment is going to be for 24 weeks and be followed by transitional period, which is for maximal 4 weeks. After that, duration of open label treatment is going to be conducted for 24 weeks. And an extension treatment will be continued until the approval or termination.
  Interventions: Drug: KW-0761 0.3 mg/kg IV
- Placebo (saline) (Placebo Comparator): Intravenous injection every 12 weeks. Duration of double-blind treatment is going to be for 24 weeks and be followed by transitional period, which is for maximal 4 weeks. After that, duration of open label treatment is going to be conducted for 24 weeks. And an extension treatment will be continued until the approval or termination.
  Interventions: Drug: Placebo (saline)

INTERVENTIONS:
Drug: KW-0761 0.3 mg/kg IV — Intravenous injection every 12 weeks.
  Arms: KW-0761 0.3 mg/kg IV
Drug: Placebo (saline) — Intravenous injection every 12 weeks.
  Arms: Placebo (saline)

SUMMARY:
The objective of this study is to assess the efficacy and safety of KW-0761 after intravenous injections in subjects with HTLV-1 associated myelopathy (HAM) in Japan.

DETAILED DESCRIPTION:
The effects of KW-0761 (0.3 mg/kg) on the Osame's motor disability score (OMDS) of subjects with HTLV-1 associated myelopathy (HAM).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent to participate in the study
2. Diagnosis as HAM according to the second edition of HAM Treatment Manual
3. At least 1-year history of HAM
4. Ongoing medication*1 for HAM, with no changes in 3 months before enrollment; or inadequate response or intolerance to prior medication,*2 which must have been discontinued for at least 3 months before enrollment. Subjects on maintenance therapy with steroids must have been receiving ≤ 10 mg/day prednisolone equivalent continuously for at least 3 months before enrollment.

   * 1 Steroids, salazosulfapyridine, or ≥ 1.5 g/day vitamin C
   * 2 Steroids, Interferon-α, salazosulfapyridine, or ≥ 1.5 g/day vitamin C
5. No change in the degree of motor dysfunction for at least 3 months before the date of screening, as judged by the investigator or subinvestigator
6. A OMDS of ≥3 at screening and able to walk ≥10 m at screening (use of a single cane or double canes is allowed)

Exclusion Criteria:

1. Any of the following significant concomitant diseases:

   Type 1 diabetes mellitus, Poorly controlled type 2 diabetes mellitus (HbA1c (NGSP) > 8.5%), Congestive heart failure (Class II to IV of the New York Heart Association Functional Classification), Myocardial infarction within 1 year before enrollment, Unstable angina within 1 year before enrollment, Poorly controlled hypertension (systolic blood pressure > 150 mm Hg and diastolic blood pressure > 90 mm Hg at screening), Sever chronic lung disease requiring oxygen therapy, Multiple sclerosis or any other demyelinating disease, Epilepsy requiring treatment with antiepileptics (with the exception of epilepsy controlled by antiepileptics, with no occurrence of seizures for at least 3 years before informed consent), and Active malignancy (including ATL); or onset of malignancy or previous treatment for malignancy (with the exception of resected or surgically cured intraepithelial carcinoma of the uterine cervix, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or ductal breast carcinoma) within 5 years before informed consent
2. Active infection
3. Concurrent spinal cord compression lesion (e.g., cervical spine diseases, disk herniation, or ossification of the ligamentum flavum) , with the exception of conditions that would not affect efficacy evaluation in the study, as judged by the investigator or subinvestigator
4. Concurrent dementia
5. Concurrent psychiatric disorder, with the exception of conditions that would not affect obtaining informed consent or efficacy evaluation in the study, as judged by the investigator or subinvestigator
6. History of or current alcohol or drug dependence
7. Planned surgery during the study period
8. Any other conditions unsuitable for participation in the study in the opinion of the investigator or subinvestigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Improvement in Osame's motor disability score | At week 4, 8 and 12 after second injection

SECONDARY OUTCOMES:
HTLV-1 Proviral load in peripheral blood | Pre-dose, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 weeks post-dose
Mean of twice 10 m walking time | Pre-dose, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 weeks post-dose
Modified Ashworth Scale | Pre-dose, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 weeks post-dose
Evaluation of Clinical Global Impression (CGI-I) | Pre-dose, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 weeks post-dose
Evaluation of Clinical Global Impression (VAS) | Pre-dose, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 weeks post-dose
Evaluation of Urinary dysfunction (OABSS) | Pre-dose, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 weeks post-dose
Evaluation of Urinary dysfunction (I-PSS) | Pre-dose, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 weeks post-dose
Evaluation of sensory dysfunction (numbness in the lower limbs (VAS)) | Pre-dose, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 weeks post-dose
Evaluation of sensory dysfunction (Pain in the lower limbs (VAS)) | Pre-dose, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 weeks post-dose
Neopterine Concentration in CSF | At week 12

CONTACTS AND LOCATIONS:
Locations (16):
- Japan (16):
  - Nagoya University Hosipital, Nagoya, Aichi-ken
  - Ehime University Hospital, Tone, Ehime
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Hospital of the University of Occupational and Environmental Health, Japan, Kitakyushu, Fukuoka
  - Kagoshima City Hospital, Kagoshima, Kagoshima-ken
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Tohoku University Hosipital, Sendai, Miyagi
  - Fujimoto General Hospital, Miyakonojō, Miyazaki
  - Oita Prefectural Hospital, Ōita, Oita Prefecture
  - National Hospital Organization Okinawa National Hospital, Ginowan, Okinawa
  - University of the Ryukyus Hospital, Nakagami, Okinawa
  - Kansai Medical University Hosipital, Hirakata, Osaka
  - University Hosipital, Kyoto Prefectural University of Medicine, Kyoto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sato T, Nagai M, Watanabe O, Misu T, Takenouchi N, Ohkubo R, Ishihara S, Tsuboi Y, Katsuno M, Nakagawa M, Matsushita T, Aso Y, Matsuura E, Tokashiki T, Mukaino A, Adachi H, Nakanishi K, Yamaguchi Y, Yamaguchi S, Yamano Y. Multicenter, randomized, double-blind, placebo-controlled phase 3 study of mogamulizumab with open-label extension study in a minimum number of patients with human T-cell leukemia virus type-1-associated myelopathy. J Neurol. 2024 Jun;271(6):3471-3485. doi: 10.1007/s00415-024-12239-x. Epub 2024 Mar 2. PMID 38430272